CLINICAL TRIAL: NCT02671786
Title: Community Based Management of Severe Malnutrition in Under 5 Children in Tribal Area of Melghat, Maharashtra- Cluster Randomized Control Field Trial
Brief Title: Community Based Management of Severe Malnutrition in Tribal Area of Melghat- Cluster Randomized Control Field Trial
Acronym: SAMMAN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MAHAN Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT-2 SAMMAN
Record Dates: First submitted 2016-01-10; First posted 2016-02-02 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Child Nutrition Disorders; Malnutrition
Keywords: Severe Acute Malnutrition; Severe Underweight; IAP Grade III-IV; Severe Stunting; Village Health Workers; MAHAN RUTF & MAHAN Vit-Mim mix
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition; Severe Acute Malnutrition; Thinness; Growth Disorders

ARMS (2):
- Intervention Arm (Experimental): Intervention area: Provision of community based health care to severely malnourished children 6 months age in 16 tribal villages by trained semi-literate village health workers.
  1. Treatment of severely malnourished children through MAHAN RUTF & MAHAN Vit-Min mix
  2. Growth monitoring of all children below the age of 5 years
  3. Treatment of associated diseases like Diarrhea, Pneumonia, Malaria, etc.
  4. Management of resistant or relapsed severely malnourished cases by pediatrician.
  5. Intensive behavior change communication of parents of children below the age of 5 years for proper nutrition.
  Dose: 46 gms of proteins/kg/day & 100170 calories/kg/day with gradual escalation with micro nutrient supplementation Route: Oral Frequency: 4 times a day Duration: 12 weeks
  Interventions: Other: MAHAN RUTF & MAHAN Vit-Min mix
- Control Arm (No Intervention): Control area: In control area, the V.H.W. and supervisor records weight of all under 5 children. They also collect data related to birth, deaths and verbal autopsy.

INTERVENTIONS:
Other: MAHAN RUTF & MAHAN Vit-Min mix — MAHAN RUTF dishes are locally prepared by local tribal women and each packet of RUTF provides 500-550 calories & 15-17 gms of proteins.
  Arms: Intervention Arm

SUMMARY:
Provision of community based health care to severely malnourished children (Age group: 6 months through 5 years) in 16 tribal villages by trained semi-literate village health workers.

1. Treatment of severely malnourished children.
2. Growth monitoring of all children below the age of 5 years.
3. Treatment of associated diseases like Diarrhea, Pneumonia, Malaria, etc.
4. Management of resistant or relapsed severely malnourished cases by pediatrician.
5. Intensive behavior change communication of parents of children below the age of 5 years for proper nutrition.

DETAILED DESCRIPTION:
1. Title of project: SAMMAN- Community based management of severe malnutrition in under 5 children in tribal area of Melghat region

2. Name of Institution: MAHAN Trust, Address: Mahatma Gandhi Tribal Hospital, Karmagram . Utavali, tehsil- Dharni, Melghat (Amaravati)

3. Objectives -

1. To reduce the child mortality (in the age of group of 6 months to 5 years) due to severe malnutrition in tribal area of Melghat by 35% in usual residents population of 15000 (from 16 villages) over a period of 3 years.
2. To reduce the prevalence of severe malnutrition (in the age of group of 6 months to 5 years) by at least 35% in usual residents population of 15000 from 16 villages in tribal area of Melghat over a period of 3 years.
3. To achieve Case fatality rate of 2 % of treated severely malnourished children.
4. Need and rational of the project :

   Melghat is a hilly difficult to approach tribal forest terrain in Amaravati district of Maharashtra, India . Population is 2,80,000 & 75% of them are tribal. Most of the tribal (>90 %) are farmers or laborers, living below poverty line(>75%) & very hard life in huts without electricity (>90%) & illiterate (>50%). Medical facilities are worst in Melghat as compared to rest of Maharashtra. A detailed study conducted by MAHAN showed that more than 20% of tribal children are severely malnourished and the under 5 children mortality rate is more than 100 per 1000 live births due to lack of proper nutrition, medical facilities, superstitions & reluctance for hospitalization of severely malnourished children. There is an immediate need to fight severe malnutrition in children between the ages of 6 months to 5 years. This project is being implemented as a pilot project in 16 villages of Melghat which has potential for replication in all tribal and rural part of India.
5. Methodology Study design: The study is a cluster randomized parallel group controlled field trial Study area: 35 tribal villages selected from 5 clusters of Melghat by lottery method divided into intervention and control area.

   Sample size - 1500 severely malnourished children from intervention and control area each.
6. Intervention:

Provision of community based health care to severely malnourished children (Age group: 6 months through 5 years) in 16 tribal villages by trained semi-literate village health workers.

1. Treatment of severely malnourished children .
2. Growth monitoring of all children below the age of 5 years.
3. Treatment of associated diseases like Diarrhea, Pneumonia, Malaria, etc.
4. Management of resistant or relapsed severely malnourished cases by pediatrician.
5. Intensive behavior change communication of parents of children below the age of 5 years for proper nutrition.

   6. Duration: 5 years (May 2011 to September 2015)

   7. Monitoring indicators for the outcome objectives:

Primary outcomes

1. Prevalence of severe malnutrition (Severe Acute Malnutrition; Severe Underweight and Indian Academy of Pediatrician (IAP) Grade III, IV)
2. No. of child deaths due to severe malnutrition
3. Case fatality rate of treated severely malnourished children

   The secondary outcomes
4. Child mortality rate between 6 to 60 months age group

   The secondary outcomes
5. Child mortality rate between 6 to 60 months age group

8. Scope & end result expected of project

1. Lives of 1500 severely malnourished children from Melghat will be saved.
2. This model of community based management of severe malnourished children using RUTF prepared by local tribal females from local produce will have better socio-cultural acceptance by parents, and will be palatable for children, hence will be more effective.
3. It will also be useful in long term for preventing recurrences and roll back cases as parents awareness will be improved with behavior change communication.
4. Based on this study, national and international policies related to community based management of severely malnourished children may be framed.
5. It will be a step towards fulfillment of fundamental rights of children guaranteed by constitution of India.

ELIGIBILITY:
Inclusion Criteria:

* Children suffering from severe malnutrition as per weight for height criteria (WHO), weight for age criteria (WHO), MUAC (WHO), IAP grade III & IV. Defacto method.

Exclusion Criteria:

* Children who have failed in appetite test and cannot tolerate oral F75 food. Also,
* Parents, guardian refuse to give consent.

Ages: 6 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 824 (Actual)
Dates: Start 2011-05; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Recovery rate of SAM (Severe Acute Malnutrition), SUW (Severe Underweight) and IAP Grade III,IV | At the end of therapeutic cycle of 3 months
Case fatality rate of treated severely malnourished children | At the end of therapeutic cycle of 3 months
Prevalence of severe malnutrition (SAM, SUW, IAP Grade III,IV) | Over the period of 3 years

SECONDARY OUTCOMES:
Child mortality rate ( 6 months to 60 months age group) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Vibhawari Dani, MBBS; MD, Principal Investigator — Research Director
Locations (1):
- MAHAN Trust, Melghat (Dharni), Amravati, Maharashtra, India

REFERENCES:
- [Background] Management of Severe Under Nutrition, A Manual for Physicians and Other Health Workers. Geneva: WHO; 1999.
- [Background] Pelletier DL, Frongillo EA Jr, Schroeder DG, Habicht JP. The effects of malnutrition on child mortality in developing countries. Bull World Health Organ. 1995;73(4):443-8. PMID 7554015
- [Background] Meshram II, Arlappa N, Balakrishna N, Laxmaiah A, Mallikarjun Rao K, Gal Reddy Ch, Ravindranath M, Sharad Kumar S, Brahmam GN. Prevalence and determinants of undernutrition and its trends among pre-school tribal children of Maharashtra State, India. J Trop Pediatr. 2012 Apr;58(2):125-32. doi: 10.1093/tropej/fmr035. Epub 2011 May 4. PMID 21543411
- [Background] Dani V, Satav A, Pendharkar J, Ughade S, Jain D, Adhav A et al. Prevalence of under nutrition in under-five tribal children of Melghat: A community based cross sectional study in Central India, Clinical Epidemiology and Global Health 2014 Sept, I-8
- [Background] Amsalu S, Tigabu Z. Risk factors for severe acute malnutrition in children under the age of five: A case-control study. Ethiop J Health Dev. 2008; 22(1): 21-5.
- [Background] Ashworth A. Efficacy and effectiveness of community-based treatment of severe malnutrition. Food Nutr Bull. 2006 Sep;27(3 Suppl):S24-48. doi: 10.1177/15648265060273S303. PMID 17076212
- [Background] WHO/UNICEF/WFP/SCN Joint statement. Community-based management of severe malnutrition. Geneva, New York, Rome, 2007
- [Background] Manary MJ, Ndkeha MJ, Ashorn P, Maleta K, Briend A. Home based therapy for severe malnutrition with ready-to-use food. Arch Dis Child. 2004 Jun;89(6):557-61. doi: 10.1136/adc.2003.034306. PMID 15155403
- [Background] Schoonees A, Lombard M, Musekiwa A, Nel E, Volmink J. Ready-to-use therapeutic food for home-based treatment of severe acute malnutrition in children from six months to five years of age. Cochrane Database Syst Rev. 2013 Jun 6;2013(6):CD009000. doi: 10.1002/14651858.CD009000.pub2. PMID 23744450
- [Background] Bergeron G, Castleman T. Program responses to acute and chronic malnutrition: divergences and convergences. Adv Nutr. 2012 Mar 1;3(2):242-9. doi: 10.3945/an.111.001263. PMID 22516735
- [Background] Ashworth A., Community-Based Rehabilitation of Severely Malnourished Children: a Review of Successful Programmes. London School of Hygiene and Tropical Medicine. Report. 2001
- [Background] Dasgupta R, Sinha D, Yumnam V. Programmatic response to malnutrition in India, room for more than one elephant. Indian Pediatr. 2014 Nov;51(11):863-8. doi: 10.1007/s13312-014-0518-5. PMID 25432212
- [Background] Dasgupta R, Ahuja S, Yumnam V. Can nutrition rehabilitation centers address severe malnutrition in India? Indian Pediatr. 2014 Feb;51(2):95-9. doi: 10.1007/s13312-014-0341-z. PMID 24632690
- [Background] Rogers BL , Rajabiun S, Levinson J, Tucker K. Reducing Chronic Malnutrition in Peru: A Proposed National Strategy
- [Background] READY-TO-USE THERAPEUTIC FOOD FOR CHILDREN WITH SEVERE ACUTE MALNUTRITION- A position paper by UNICEF
- [Background] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- Available data/document: Pilot Study Research Paper — http://www.worldwidejournals.com/ijar/file.php?val=April_2015_1427896145__152.pdf